CLINICAL TRIAL: NCT03242174
Title: Health Behaviors in Pregnancy
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2017-036
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prenatal Care Late; Pregnancy Related; Lifestyle

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional Obstetrical Prenatal Care: Pregnant women receiving traditional obstetrical prenatal care and delivering in a hospital will be offered the Health Behavior questionnaire packet at third trimester prenatal appointment
  Interventions: Other: Health Behavior Questionnaire Packet
- Prenatal Care from Midwife: Pregnant women receiving prenatal care from a midwife and delivering at the birth center will be offered the Health Behavior questionnaire packet at third trimester prenatal appointment
  Interventions: Other: Health Behavior Questionnaire Packet

INTERVENTIONS:
Other: Health Behavior Questionnaire Packet — Any pregnant woman offered the questionnaire at her prenatal appointment in the third trimester can complete

SUMMARY:
To assess health and lifestyle behavior of pregnant women in Baton Rouge including women receiving traditional obstetrical prenatal care and delivering in a hospital and those receiving prenatal care from a midwife and delivering at the birth center.

DETAILED DESCRIPTION:
It is of scientific interest to learn what the health and lifestyle behaviors are for women receiving prenatal care in a non-traditional birth center and the impact of these behaviors on pregnancy and birth outcomes.Participants will be offered a questionnaire packet to complete at a prenatal appointment in the third trimester of pregnancy by their obstetrical prenatal care provider. The questionnaire packet will take approximately 10-15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester of pregnancy ≥ 28 weeks GA

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women in the third trimester of pregnancy ≥ 28 weeks GA will be offered the opportunity to participate in this study at the time of a prenatal appointment ≥ 28 weeks GA
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Eating Habits | 1 Day
  Eating Habits assessed by Eating Habits Questionnaire
Eating Habits | 1 Day
  Eating Habits assessed by Rapid Eating Assessment for Participants-Shortened Version
Mindful Eating | 1 Day
  Mindful Eating assessed by Mindful Eating Questionnaire
Physical Activity | 1 Day
  Physical Activity assessed by Nurses Health Study II Physical Activity Questionnaire
Frequency of Weighing | 1 Day
  Frequency of Weighing by Frequency of Weighing Questionnaire
Sedentary Behavior | 1 Day
  Sedentary Behavior by Sedentary Behavior Questionnaire
Functional health and well-being | 1 Day
  Quality of life measure that assesses functional health and well-being from the participant's point of view by 12 Item Short Form Health Survey by RAND
Sleep Habits | 1 Day
  Sleep Habits by Sleep Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No